CLINICAL TRIAL: NCT05973006
Title: A Phase 3, Randomized, Double-Blinded Study to Evaluate the Safety and Immunogenicity of Omicron Subvariant and Bivalent SARS-CoV-2 rS Vaccines in Adolescents Previously Vaccinated With mRNA COVID-19 Vaccines
Brief Title: Phase 3 Adolescent Study for SARS-CoV-2 rS Variant Vaccines
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019nCoV-314
Record Dates: First submitted 2023-07-31; First posted 2023-08-02 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group-A NVX-CoV2601 (Experimental): The Monovalent NVX-CoV2601 of 5 μg of antigen with 50 μg of Matrix-M adjuvant
  Interventions: Biological: NVX-CoV2601 co-formulated Omicron XBB.1.5 SARS-CoV-2 rS vaccine
- Group-B Bivalent NVX CoV2373 + NVX CoV2601 (Active Comparator): The Bivalent NVX CoV2373 + NVX CoV2601 of 5 μg of each antigen with a total of 50 μg of Matrix-M adjuvant
  Interventions: Biological: Prototype/XBB.1.5 Bivalent Vaccine (5 µg)

INTERVENTIONS:
Biological: NVX-CoV2601 co-formulated Omicron XBB.1.5 SARS-CoV-2 rS vaccine — Coformulated Omicron XBB.1.5 SARS-CoV-2 rS vaccine with Matrix-M adjuvant: supplied as a solution for preparation for injection, at a concentration of 10 µg antigen and 100 µg adjuvant per mL. All injections will be administered in a 0.5 mL injection volume at a dose of 5 µg antigen with 50 µg Matrix-M adjuvant.
  Other Names: NVX-CoV2601
  Arms: Group-A NVX-CoV2601
Biological: Prototype/XBB.1.5 Bivalent Vaccine (5 µg) — A site-mixed bivalent vaccine prepared by combining 0.25 mL of NVX-CoV2373 and 0.25 mL NVX-CoV2601. All injections will be administered in a 0.5 mL injection volume at a dose of 5 µg total antigen (2.5 µg prototype antigen + 2.5 µg Omicron XBB.1.5 antigen) with 50 µg Matrix-M adjuvant.
  Other Names: Omicron XBB.1.5 (sub-variant)SARS-CoV-2 rS /Matrix-M Adjuvant
  Arms: Group-B Bivalent NVX CoV2373 + NVX CoV2601

SUMMARY:
This study is a large-scale investigation (Phase 3) into a new booster shot designed specifically for teenagers. The booster targets a particular variant of COVID-19, Omicron XBB.1.5. The main focus is on safety: researchers want to see if this new booster is safe for teenagers who have already received two doses of the Pfizer or Moderna mRNA COVID-19 vaccines. To ensure a fair comparison, the study will use a double-blind approach. This means two groups of teenagers will receive booster shots, but neither the teenagers nor the researchers giving the shots will know beforehand which version of the booster each person gets. The study will also assess how well the body fights the virus after the booster shot.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blinded study to evaluate the safety and immunogenicity of booster doses of Omicron subvariant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccines (SARS-CoV-2 rS) adjuvanted with Matrix-M™ adjuvant (NVX-CoV2601 [Omicron XBB.1.5]) and bivalent (NVX-CoV2373 [prototype] + NVX CoV2601) in previously vaccinated adolescent participants ≥ 12 to < 18 years of age.

Approximately 400 adolescents who have received a regimen of ≥ 2 doses of the Moderna and/or Pfizer-BioNTech monovalent and/or bivalent COVID-19 vaccines ≥ 90 days previously will be randomized 1:1 to Group A or Group B:

* Group A: 1 dose of NVX-CoV2601 (1 on Day 0)
* Group B: 1 dose of bivalent NVX-CoV2373 + NVX-CoV2601 (1 on Day 0) All participants will remain on study for immunogenicity and safety data collection through Day 180.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents ≥ 12 to < 18 years of age at screening
2. Participant and parent(s)/caregiver(s) or legally acceptable representative willing and able to give in-formed consent and assent, as required, prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or post-menopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.
6. Have previously received ≥ 2 doses of the Moderna and/or Pfizer-BioNTech monovalent and/or bivalent COVID-19 vaccines with the last dose having been given ≥ 90 days previously prior to study vaccination.

Exclusion Criteria:

1. Received COVID-19 vaccines other than Moderna and/or Pfizer-BioNTech in the past, inclusive of clinical trial COVID-19 vaccines.
2. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to study vaccination.
3. Received influenza vaccination within 14 days prior to study vaccination.
4. Received any vaccine ≤ 45 days prior to study vaccination, except for rabies, human papilloma virus (HPV), tetanus-diphtheria (Td), tetanus, diphtheria, and pertussis (TDaP/DTap), hepatitis B virus (HBV), and meningococcal vaccines which may be given as medically indicated.
5. Any known allergies to products contained in the investigational product.
6. Any history of anaphylaxis to any prior vaccine.
7. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.
8. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination.

   An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.
9. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination, except for rabies immunoglobulin which may be given if medically indicated.
10. Active cancer (malignancy) on therapy within 3 years prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
11. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
12. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
13. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
14. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
15. Participants with a history of myocarditis or pericarditis.
16. Respiratory symptoms in the past 3 days (ie, cough, sore throat, difficulty breathing).
17. Temperature of > 38°C within 24 hours of planned study vaccination (site measured or participant measured).
18. Blood pressure of ≥ 160/100 mmHg.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (20):
- United States (20):
  - Alfa Medical Research, Davie, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - ITB Research, Miami, Florida
  - Velocity Clinical Research, Meridian, Idaho
  - DM Clinical Research - Chicago, River Forest, Illinois
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC (AMR), Newton, Kansas
  - AMR, Wichita, Kansas
  - Velocity Clinical Research, Lafayette, Louisiana
  - Velocity Clinical Research, Vestal, New York
  - Velocity Clinical Research, Cincinnati, Ohio
  - Tekton Research, Tulsa, Oklahoma
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - DM Clinical Research, Houston, Texas
  - Medical Colleagues of Texas, LLP, Katy, Texas
  - Research Your Health, Plano, Texas
  - Tekton Research, San Antonio, Texas
  - Mountain View CCT Research, Pleasant View, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Started | 190 | 210
Completed | 187 | 201
Not Completed | 3 | 9
Not completed — Early termination | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601 | Total
Number analyzed (Participants) | 190 | 210 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.77) | 14.5 (1.65) | 14.5 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 107 | 206
  Male | 91 | 103 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 47 | 90
  Not Hispanic or Latino | 147 | 163 | 310
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 33 | 44 | 77
  White | 137 | 149 | 286
  More than one race | 9 | 10 | 19
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Participants With Solicited Local and Systemic AEs for 7 Days Following Vaccination
Description: Participants with solicited local and systemic adverse events (AEs) To assess the overall safety of 1 heterologous booster dose of NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) for 7 days following vaccination
Time Frame: Day 7
Measure: Number; unit: participants
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 190 | 210
participants
  Any Solicited AEs | 153 | 166
  Local AEs | 136 | 140
  Systemic AEs | 116 | 120

2. Primary Outcome: Participants With Unsolicited AEs Through 28 Days After Vaccination
Description: Participants with unsolicited AEs to assess the overall safety of 1 heterologous booster dose of NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) through 28 days after vaccination.
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 190 | 210
participants
  Any unsolicited TEAE through 28 days after study vaccination | 25 | 25
  Infections and infestations | 15 | 13
  Psychiatric disorders | 4 | 2
  General disorders and administration site conditions | 3 | 3
  Respiratory, thoracic and mediastinal disorders | 2 | 3
  Gastrointestinal disorders | 3 | 1
  Skin and subcutaneous tissue disorders | 2 | 1
  Injury, poisoning and procedural complications | 2 | 0
  Blood and lymphatic system disorders | 1 | 1
  Musculoskeletal and connective tissue disorders | 1 | 1
  Nervous system disorders | 0 | 1
  Metabolism and nutrition disorders | 0 | 1

3. Primary Outcome: Participants With (MAAEs) Attributed to Study Vaccine, (AESIs) (PIMMCs), Myocarditis and/or Pericarditis, and Complications Specific to COVID-19), and Serious Adverse Events (SAEs)
Description: Participants with medically attended adverse events (MAAEs) attributed to study vaccine, adverse events of special interest (AESIs) (predefined list including potential immune-mediated medical conditions (PIMMCs), myocarditis and/or pericarditis, and complications specific to COVID-19), and serious adverse events (SAEs) o assess the overall safety of 1 heterologous booster dose of NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601)through day 180 or end of study (EOS).
Time Frame: Day 180
Measure: Number; unit: participants
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 190 | 210
participants
  Any TEAEs | 25 | 25
  Any MAAEs | 16 | 12
  Any Serious TEAEs | 4 | 1

4. Primary Outcome: Immunogenicity Index- Neutralizing Antibody (NAb) Expressed as Geometric Mean Titers (GMTs) to the Omicron XBB.1.5 Strain.
Description: The neutralizing antibody (NAb) response induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the Omicron XBB.1.5 strain assessed at Day 28 following initial study vaccination.
Time Frame: Day 0 and Day 28
Population: Per Protocol Neutralization Assay Subset Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 178 | 194
geometric mean titer
  Day 0 | 208.40 [166.20 to 261.32] | 184.81 [148.86 to 229.45]
  Day 28 | 2533.08 [2107.17 to 3045.07] | 1544.61 [1314.33 to 1815.25]

5. Primary Outcome: Immunogenicity Index- The Neutralizing Antibody (NAb) Expressed as Geometric Mean Fold Rise (GMFR) to the Omicron XBB.1.5 Strain.
Description: the neutralizing antibody (NAb) response induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the Omicron XBB.1.5 strain, assessed at Day 28
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 178 | 194
geometric mean fold rise | 12.2 [9.5 to 15.5] | 8.4 [6.8 to 10.3]

6. Secondary Outcome: Neutralizing Antibody (NAb) Expressed as Geometric Mean Titers (GMTs) to the Omicron XBB.1.5 Strain.
Description: the neutralizing antibody NAb response induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the Omicron XBB.1.5 strain over time. at relevant time points.
Time Frame: Day 0 to Day 180
Population: Per Protocol Neutralization Assay Subset Population
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 180 | 196
geometric mean titer
  Day 0 | 204.98 [163.68 to 256.69] | 183.37 [147.82 to 227.47]
  Day 28: number analyzed (Participants) | 178 | 194
  Day 28 | 2533.08 [2107.17 to 3045.07] | 1544.61 [1314.33 to 1815.25]
  Day 90: number analyzed (Participants) | 177 | 186
  Day 90 | 1816.50 [1505.62 to 2191.56] | 1171.90 [997.69 to 1376.52]
  Day 180: number analyzed (Participants) | 168 | 177
  Day 180 | 1369.61 [1128.29 to 1662.53] | 866.10 [733.49 to 1022.67]

7. Secondary Outcome: Neutralizing Antibody (NAb) Expressed as Geometric Mean Fold Rise (GMFR) to the Omicron XBB.1.5 Strain.
Description: as for outcome 6
Time Frame: Day 28 to Day 180
Population: Per Protocol Neutralization Assay Subset
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold rise
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 180 | 196
geometric mean fold rise
  Day 28: number analyzed (Participants) | 178 | 194
  Day 28 | 12.2 [9.5 to 15.5] | 8.4 [6.8 to 10.3]
  Day 90 | 8.6 [6.7 to 11.1] | 6.2 [5.0 to 7.7]
  Day 180 | 6.0 [4.7 to 7.8] | 4.7 [3.7 to 5.9]

8. Secondary Outcome: IgG Geometric Mean ELISA (Enzyme-linked Immunosorbent Assay) Units (GMEUs) to the Omicron XBB.1.5 S Protein.
Description: The immunoglobulin G (IgG) antibody levels induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the Omicron XBB.1.5 strain over time.at relevant time points.
Time Frame: Day 0 to Day 180
Population: Per Protocol Anti-S Protein IgG Serology Subset Population
Measure: Geometric Mean (95% Confidence Interval); unit: Elisa Units per mL
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 180 | 196
Elisa Units per mL
  Day 0 | 38825.1 [33160.1 to 45457.9] | 32881.9 [28434.7 to 38024.7]
  Day 28: number analyzed (Participants) | 178 | 194
  Day 28 | 150232.9 [132853.6 to 169885.6] | 113031.9 [101227.0 to 126213.4]
  Day 90: number analyzed (Participants) | 177 | 186
  Day 90 | 110091.1 [96294.7 to 125864.3] | 87102.4 [77115.6 to 98382.6]
  Day 180 | 77149.8 [68110.5 to 87388.8] | 61647.7 [55459.2 to 68526.7]

9. Secondary Outcome: NAb(Neutralizing Antibody Titers) Levels Are Measured to the Ancestral (Wuhan) Strain .
Description: The NAb antibody responses induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the ancestral (Wuhan) strain at relevant time points .
Time Frame: Day 0 to 180
Population: Per Protocol Neutralization Assay Subset
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 180 | 196
geometric mean titer
  Day 0 | 1321.00 [1123.04 to 1553.87] | 1197.59 [1029.90 to 1392.58]
  Day 28: number analyzed (Participants) | 178 | 194
  Day 28 | 3510.84 [3099.99 to 3976.14] | 2803.80 [2453.96 to 3203.51]
  Day 90 | 3381.08 [2991.33 to 3821.62] | 2924.82 [2581.96 to 3313.23]
  Day 180 | 2663.87 [2334.49 to 3039.72] | 2357.51 [2095.11 to 2652.77]

10. Secondary Outcome: Serum IgG GMEUs Levels Are Measured to the Ancestral (Wuhan) Strain .
Description: The serum IgG antibody responses induced by NVX CoV2601 and the bivalent vaccine (NVX CoV2373 + NVX-CoV2601) against the ancestral (Wuhan) strain at relevant time points.
Time Frame: Day 0 to Day 180
Population: Per Protocol Anti-S Protein IgG Serology Subset
Measure: Geometric Mean (95% Confidence Interval); unit: Elisa Units per mL
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
Number analyzed (Participants) | 180 | 196
Elisa Units per mL
  Day 0 | 71388.4 [62262.8 to 81851.6] | 61296.9 [53962.1 to 69628.5]
  Day 28 | 181736.6 [162092.7 to 203761.1] | 157077.8 [141109.2 to 174853.4]
  Day 90 | 142032.4 [124824.9 to 161611.9] | 130155.1 [116798.0 to 145039.8]
  Day 180 | 104890.2 [93135.9 to 118128.0] | 94026.0 [84606.1 to 104494.8]

ADVERSE EVENTS:
Time Frame: 180 Days
Arm/Group | Group-A NVX-CoV2601 | Group-B Bivalent NVX CoV2373 + NVX CoV2601
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/210
Serious Adverse Events (participants affected / at risk) | 7/190 | 1/210
Other Adverse Events (participants affected / at risk) | 10/190 | 4/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A NVX-CoV2601 (N=190) | Group-B Bivalent NVX CoV2373 + NVX CoV2601 (N=210)
Adjustment disorder with anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A NVX-CoV2601 (N=190) | Group-B Bivalent NVX CoV2373 + NVX CoV2601 (N=210)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT05973006/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05973006/SAP_001.pdf